CLINICAL TRIAL: NCT06861699
Title: Kan Akımı Kısıtlayıcı Egzersizin Kas Mekanikleri Üzerine Akur Etkisi
Brief Title: Blood Flow Technique Effect on the Muscle Mechanics
Status: Not yet recruiting | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Melis Destan, Assistant Professor, Okan University
Other Study IDs: 2024-34
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Biceps; Muscle Rigidity
MeSH Terms: conditions — Muscle Rigidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- progressive resistance exercise group with bfr (%80): Participants in this group will perform progressive resistance exercises with 80% blood flow restriction (BFR) exposure, while muscle mechanical properties will be monitored and recorded during the process.
- progressive resistance exercise group with bfr (%20): Participants in this group will perform progressive resistance exercises with 20% blood flow restriction (BFR) exposure, while muscle mechanical properties will be monitored and recorded during the process.
- Non-Blood Flow Restriction Group: Participants in this group will perform progressive resistance exercises without applying the blood flow restriction (BFR) technique, while muscle mechanical properties will be monitored and recorded during the process."

SUMMARY:
This study will be a study in which we take measurements with the myotonPRO device to determine whether the resistant exercises performed without the blood flow restrictive technique and with the blood flow restrictive technique affect the biceps muscle of the participants, who were divided into groups by randomization method after determining the 1 max repetition you can lift.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy male or female volunteer between 18 and 35 (who has not participated in any resistance training program for at least 6 months).
* Being right-hand dominant according to the results of the Edinburgh Handedness Inventory.

Exclusion Criteria:

* Having a history of biceps musculoskeletal injury.
* Having any condition that prevents participation in resistance exercise.
* Having cardiovascular disease.
* Using medication for blood pressure control.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: generally college students
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
muscle mechanics test | Single assessment at baseline and one, two and three days after with measurement